CLINICAL TRIAL: NCT01642628
Title: The Effect of Pre-Operative Education and Self-Reflection on Anxiety, Body Image, Depression and Emotional Well-Being of Women Undergoing Mastectomy
Brief Title: The Effect of Mirror Education for Women Undergoing Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Memorial Hermann Health System (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Wyona M. Freysteinson, PhD, MN, Assistant Professor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17006
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Emotional Distress; Anxiety; Depression
Keywords: Mirror; Body Image; Mastectomy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Body Image/Mirror Education (Experimental): Participants in the mirror arm will receive a mirror and mirror viewing education from oncology nurse navigators.
  Interventions: Other: Mirror Education
- Standard Care (No Intervention): Patients allocated to the control group will receive the usual pre and post-op standard care that does not include the use or discussion of mirrors.

INTERVENTIONS:
Other: Mirror Education — Patients allocated to the experimental group will be given a small hand-held mirror and structured mirror viewing education verbally. In addition, they will receive a mirror viewing handout. This intervention will be given prior to mastectomy surgery. In addition, participants will receive all other standard care.
  Other Names: Experimental group
  Arms: Body Image/Mirror Education

SUMMARY:
Intuitively, the investigators surmise the initial and subsequent viewing of a breast site following mastectomy may be traumatic. A qualitative study on the experience of viewing self in the mirror for a woman who has had a mastectomy has confirmed the experience is unique for each individual, and may well be difficult. This research study aims to determine if these difficult moments may be buffered by a mirror intervention providing women who are scheduled for a mastectomy with a hand held mirror, instructions by a Oncology Nurse Navigator (ONN) on how to use the mirror in initial and subsequent dressing changes, and offering to discuss any concerns or questions.

The purpose of this study is to evaluate the feasibility of a nursing mirror educational intervention and determine if it is of potential value for women scheduled for a mastectomy. Results from this pilot study will help determine whether the research design, setting, sample, instruments, data collection and data analysis are appropriate and practical for a larger study.

Hypothesis

Women, ages 18 and over, who have had a mastectomy, and receive a planned pre-operative education and self-reflection intervention will have relatively improved anxiety, body image, depression and emotional well-being scores one to three weeks post-operatively as compared to those who received usual care.

DETAILED DESCRIPTION:
The literature suggests women view the mastectomy site in a mirror post-operatively because they 1) are curious as to what their changed body looks like 2) need to do wound care and 3) want to keep up personal appearances. Regardless of the reason a women may choose to view self, viewing the post-operative site may be emotionally difficult. To confound the issue, the literature also suggests that there are few mirrors available in hospitals, clinics and physician offices. As such, women who have had a mastectomy may be unable to choose to view self in a mirror at any time, including during initial and/or subsequent dressing changes, with the support of a health care professional. The word mirror is seldom if ever discussed, and mirrors are seldom, if ever, offered to women who have had a mastectomy.

As such, 20 women will be recruited (ten in each group)by ONNs. ONNs will give potential participants the standardized description of the study and obtain consent. After participant randomization to either interventional or control groups, ONNs will give participants in the research group a handheld mirror and a handout on mirrors and mirror viewing. ONN's will review each element of the handout with the participants. ONN's will provide emotional support as appropriate for any participant who may have concerns, fears, or questions concerning the mirror. ONNs will also proceed with usual pre-operative education.

Participants in the control group will receive usual pre-operative education. Usual pre-operative education consists of a face-to-face pre-operative appointment with the ONN. The ONN provides education about the upcoming surgery, post-operative procedures, and breast cancer support resources.

Participants will be phoned post-operatively to set up a meeting one to three weeks post-operatively to re-administer the written instruments and, in addition, administer a written structured questionnaire on the subjects' use of the mirror.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for breast cancer surgery
* Surgery to result in mastectomy where at least one entire breast is removed
* Speak, read, and understand English

Exclusion Criteria:

* Patients having a guardian that is responsible for medical decisions.
* Patients reporting a diagnosis of body dysmorphic disorder
* Patients who have undergone previous breast cancer surgery
* Patients undergoing breast reconstruction other than placement of implant(s)or tissue expander(s).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Emotional well-being | Change from pre-operative baseline up to three weeks post-operatively
  Emotional well-being will be measured using MOS 36-Item Short Form Survey (SF-36) emotional well-being subscale and Functional Assessment of Cancer Therapies (FACT) emotional well-being scale.

SECONDARY OUTCOMES:
Body image | Change from pre-operative baseline up to three weeks post-operatively
  Body image will be measured using the Body Image Scale (BIS).
Anxiety | Change from pre-operative baseline up to three weeks post-operatively
  Anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS).
Depression | Change from pre-operative baseline up to three weeks post-operatively
  Depression will be measured using the HADS.
Use of mirrors | Up to three weeks post-operatively
  Use of mirrors will be measured using a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Wyona M. Freysteinson, PhD, MN, Principal Investigator — Texas Woman's University
Locations (2):
- United States (2):
  - Memorial Hermann Healthcare System, Houston, Texas
  - Texas Woman's University, Houston, Texas

REFERENCES:
- [Background] Freysteinson WM, Deutsch AS, Lewis C, Sisk A, Wuest L, Cesario SK. The experience of viewing oneself in the mirror after a mastectomy. Oncol Nurs Forum. 2012 Jul;39(4):361-9. doi: 10.1188/12.ONF.361-369. PMID 22750894